CLINICAL TRIAL: NCT02948556
Title: ME/CFS: Activity Patterns and Autonomic Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01NR015850-01A1 (NIH)
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic fatigue syndrome: Participants with chronic fatigue syndrome

SUMMARY:
The purpose of this study is to identify daily activity patterns, negative life events and autonomic abnormalities that may be related to non-improvement in myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). For both naturalistic studies and behavioral intervention trials, roughly 50% of patients report worsening or unchanged illness. The proposed four year study would be the first to look at the relation between illness non-improvement, patient activities at home and autonomic function. Our long-range goal is to identify physiological signals and activity patterns that predict non-improvement and relapse and develop a self-management program that prescribes improvement-linked behaviors and discourages non-improvement activities.

DETAILED DESCRIPTION:
Given the enduring debilitation and poor quality of life in ME/CFS, this study proposes to identify important activity patterns (e.g., push-crash), negative life events and autonomic dysfunction that may be associated with non-improvement. This will be accomplished with weekly online diaries, objective measures (actigraphy, heart rate monitors) and semi-structured phone interviews. Non-improvement is a rarely studied, but commonly reported outcome in this illness. For both naturalistic studies and behavioral intervention trials, roughly 50% of ME/CFS patients report worsening or unchanged illness. Also, the patient's self-management efforts may (paradoxically) produce symptom worsening and contribute to illness non-improvement. Non-improvement may also have biological relevance because activity limitations and sleep disruption in ME/CFS have both been associated with autonomic dysregulation (reduced heart rate variability). This (R01) prospective observational six month study of both daily and weekly in vivo assessments would be the first to look at non-improvement in relation to ongoing patient activities and autonomic function.

Specific Aim 1: To assess the relation between non-improvement and prospectively assessed activity patterns and life events. Hypothesis 1: Non-improvement will be significantly associated with these dimensional variables: (a) illness-exacerbating activity patterns (e.g., "push-crash") reported on home web diaries; (b) daily hassles assessed in web diaries; and (c) negative life events reported in phone interviews.

Specific Aim 2: To assess the relation between improvement and prospectively assessed activity patterns and life events. Hypothesis 2: Improvement will be significantly associated with: (a) illness-moderating activity patterns (e.g., healthy pacing) reported on home web diaries; (b) daily uplifts assessed in web diaries; and (c) positive life events assessed in phone interviews.

Specific Aim 3: To assess the relation between activity patterns and symptoms. Hypothesis 3: (a) the "push-crash" pattern will predict greater actigraphy variability and symptom variability; (b) the "limiting activity" pattern will be associated with very low actigraphy counts and high symptom severity; and (c) a healthier "pacing" pattern will be associated with moderate variability of actigraphy and symptoms.

Our secondary aim hypothesizes that autonomic dysregulation (reduced heart rate variability [HRV]) will be characteristic of both non-improvers and patients with a limiting activity pattern as compared to improvers and those with a healthy pacing pattern. The long-range goal is to develop a new self-management protocol that more clearly identifies non-improvement activities and how they can be changed. An important aspect of this new self-management protocol would be to identify early signals of impending relapse, particularly HRV status, via home-use portable devices that could be utilized by patients and their doctors as a warning to modify non-improvement activities, e.g., excessive activity or exercise, to prevent behavioral collapse into inactivity.

ELIGIBILITY:
Inclusion Criteria:

Fukuda-based ME/CFS symptoms including:

* six months of unexplained, debilitating fatigue
* 4/8 secondary symptoms impaired memory or concentration unrefreshing sleep sore throats headache muscle pain joint pain tender lymph nodes post-exertional malaise

Exclusion Criteria:

Medical: fatigue clearly attributable to self-report medical conditions.

Psychiatric any psychosis alcohol/ substance abuse within two years prior or after illness onset. depression with melancholic/psychotic features within 5 years of onset .

Two other exclusionary criteria:

* patients not dose-stabilized for at least 3 months on antidepressants ;
* patients at risk of suicide or need of urgent psychiatric treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosed chronic fatigue syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Global Impression of Change Rating | six months
  Validated Self-report rating via interview

CONTACTS AND LOCATIONS:
Overall Officials: Fred Friedberg, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Friedberg F, Adamowicz JL, Bruckenthal P, Milazzo M, Ramjan S, Zhang X, Yang J. Uplifts and hassles are related to worsening in chronic fatigue syndrome: a prospective study. J Transl Med. 2023 Aug 20;21(1):557. doi: 10.1186/s12967-023-04412-z. PMID 37598161
- [Derived] Friedberg F, Adamowicz JL, Bruckenthal P, Milazzo M, Ramjan S, Zhang X, Yang J. Uplifts and hassles are related to worsening in chronic fatigue syndrome A prospective study. Res Sq [Preprint]. 2023 May 5:rs.3.rs-2865400. doi: 10.21203/rs.3.rs-2865400/v1. PMID 37205559
- [Derived] Friedberg F, Adamowicz JL, Bruckenthal P, Milazzo M, Ramjan S, Quintana D. Nonimprovement in Chronic Fatigue Syndrome: Relation to Activity Patterns, Uplifts and Hassles, and Autonomic Dysfunction. Psychosom Med. 2022 Jul-Aug 01;84(6):669-678. doi: 10.1097/PSY.0000000000001082. Epub 2022 Apr 14. PMID 35420586